CLINICAL TRIAL: NCT06832956
Title: Efficacy and Safety of Cryoablation with Robotic Bronchoscopy System in Patients with Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professsor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBS-cryoablation
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RBS group (Experimental): Cryobiopsy with Unicorn robotic bronchoscopy system
  Interventions: Procedure: robotic bronchoscopy system

INTERVENTIONS:
Procedure: robotic bronchoscopy system — cryobiopsy with the help of RBS

SUMMARY:
The goal of this single-arm clinical trial is to evaluate the safety and efficacy of robotic bronchoscopy system (RBS)-assisted cryoablation in the treatment of primary lung cancer in adult patients (aged ≥18 years) with histologically confirmed non-resectable primary lung cancer, regardless of gender. The main questions it aims to answer are:

Does RBS-assisted cryoablation achieve a predefined target technical success rate for complete tumor ablation under imaging guidance? Is the incidence of severe procedure-related adverse events within an acceptable safety threshold ?

Participants will:

Provide written informed consent for RBS-assisted cryoablation.

Undergo pretreatment evaluations, including:

Multimodal imaging (CT/PET-CT) for tumor localization and staging. Pulmonary function tests and cardiopulmonary risk assessment. Receive RBS-guided cryoablation therapy under general anesthesia. Be monitored for intraoperative complications and postoperative adverse events for 72 hours.

Complete follow-up assessments at 1, 3, 6, and 12 months post-procedure, including:

Contrast-enhanced CT scans to evaluate local tumor control. Documentation of symptom progression and quality-of-life metrics.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years old, regardless of gender. (2) Diagnosed with peripheral lung cancer, with the maximum diameter of the tumor ≤ 3 cm and the number of tumors ≤ 3. (3) The lesion to be ablated is evaluated as suitable for bronchoscopy-guided cryoablation treatment. (4) The subject refuses or is deemed unsuitable for radiotherapy/chemotherapy, or shows no response to previous radiotherapy/chemotherapy, or experiences disease progression after radiotherapy/chemotherapy. (5) Assessed as ineligible for surgery or refuses surgery and radiotherapy, consents to receive initial ablation treatment, and signs the informed consent form.

Exclusion Criteria:

* (1) Diffuse lesions in both lungs where ablation treatment is unlikely to improve the condition. (2) Presence of hilar lymph node metastasis or extrapulmonary metastasis as indicated by examinations within 1 month before the operation (except for extrapulmonary metastasis that has been controlled by local treatment). (3) Presence of contraindications for bronchoscopy, or inability to tolerate or cooperate with bronchoscopy. (4) Severe bleeding tendency, uncorrectable coagulation dysfunction (prothrombin time > 18 s, prothrombin activity < 40%). (5) Platelet count < 70×109/L, or anticoagulant and/or antiplatelet drugs have not been discontinued for more than 1 week before ablation (except for prophylactic use of low-molecular-weight heparin before the operation). (6) Severe impairment of lung function, with maximum ventilation < 40%. (7) Concurrent with other tumors and extensive metastasis, with an expected survival period of less than 3 months. (8) Poor general condition (multiple metastases throughout the body, severe infection, high fever), infectious and radiation-induced inflammation around the lesion, obvious cachexia, severe insufficiency of vital organs, severe anemia and nutritional metabolic disorders that cannot be improved in the short term. (9) Eastern Cooperative Oncology Group (ECOG) performance status score > 2. (10) The lesion to be ablated has received radiotherapy within the past 6 months. (11) Presence of active hepatitis B, active hepatitis C, history of human immunodeficiency virus (HIV) infection (known positive for HIV 1/2 antibodies), or other active infections that may affect the patient's treatment as judged by the investigator. (12) Accompanied by epilepsy, history of mental illness or cognitive impairment. (13) Pregnant or lactating women, and male or female patients planning to conceive or become pregnant during the trial. (14) Participation in any other clinical trial within 3 months before signing the informed consent form (except for non-interventional studies). (15) Other circumstances considered inappropriate for participation in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events incidence | 1 month after procedure
  The proportion of complications related to cryoablation (such as bleeding, pneumothorax, infection, etc.) that occurred in the subjects after cryoablation treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakaji H, Niimi A, Matsuoka H, Iwata T, Cui S, Matsumoto H, Ito I, Oguma T, Otsuka K, Takeda T, Inoue H, Tajiri T, Nagasaki T, Kanemitsu Y, Chin K, Mishima M. Airway remodeling associated with cough hypersensitivity as a consequence of persistent cough: An experimental study. Respir Investig. 2016 Nov;54(6):419-427. doi: 10.1016/j.resinv.2016.06.005. Epub 2016 Jul 31. PMID 27886853